CLINICAL TRIAL: NCT00532129
Title: An Open-Label Study to Characterize the Safety and Response Rate of MabThera (Rituximab) Plus Chlorambucil in Previously Untreated Patients With CD20-Positive B-Cell Chronic Lymphocytic Leukemia
Brief Title: A Study of MabThera (Rituximab) Plus Chlorambucil in Participants With Chronic Lymphocytic Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO20927; 2007-000172-16 (EudraCT Number)
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab plus Chlorambucil (Experimental): Participants will receive combination therapy of rituximab plus chlorambucil for first 6 cycles and then chlorambucil alone for a maximum of 6 additional cycles.
  Interventions: Drug: Rituximab; Drug: Chlorambucil

INTERVENTIONS:
Drug: Rituximab — 375mg/m^2 IV on Day 1 of Cycle 1; 500mg/m^2 on Day 1 of Cycles 2-6.
  Other Names: MabThera; Rituxan
Drug: Chlorambucil — 10 mg/m^2/day PO on Days 1 to 7 of each cycle for a maximum of 12 cycles.

SUMMARY:
This single arm study will assess the safety and effect on response rate of a combination of rituximab and chlorambucil in previously untreated participants with B-cell chronic lymphocytic leukemia. Participants will receive 6 monthly cycles of combination treatment, followed by up to 6 cycles of chlorambucil alone. Rituximab will be administered on Day 1 of each cycle, at a dose of 375 milligrams per square meter (mg/m^2) intravenously (IV) in Cycle 1, and 500 mg/m^2 in subsequent cycles, and chlorambucil will be administered on Days 1-7 of each cycle at a dose of 10 mg/m^2/day per oral (PO).

ELIGIBILITY:
Inclusion Criteria:

* previously untreated participants with cluster of differentiation 20 (CD20) positive B-cell chronic lymphocytic leukemia;
* participants with progressive Binet stage B, or C requiring therapy according to National Cancer Institute (NCI) criteria;
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.

Exclusion Criteria:

* previous treatment for Chronic Lymphocytic Leukaemia (CLL);
* known concomitant hematological malignancy;
* transformation to aggressive B-cell malignancy;
* history of severe cardiac disease;
* known hypersensitivity or anaphylactic reactions to murine antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United Kingdom (11):
  - Birmingham
  - Bournemouth
  - Cambridge
  - Canterbury
  - Cottingham
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Sutton
  - Wakefield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hillmen P, Gribben JG, Follows GA, Milligan D, Sayala HA, Moreton P, Oscier DG, Dearden CE, Kennedy DB, Pettitt AR, Nathwani A, Varghese A, Cohen D, Rawstron A, Oertel S, Pocock CF. Rituximab plus chlorambucil as first-line treatment for chronic lymphocytic leukemia: Final analysis of an open-label phase II study. J Clin Oncol. 2014 Apr 20;32(12):1236-41. doi: 10.1200/JCO.2013.49.6547. Epub 2014 Mar 17. PMID 24638012

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Chlorambucil: Participants received combination therapy of rituximab plus chlorambucil for first 6 cycles (28 day cycles). Participants who did not achieve complete response (CR) after Cycle 6 then received chlorambucil alone from Cycle 7 onwards until either they achieved a CR or for a maximum of 6 additional cycles. Rituximab: 375 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 of Cycle 1; 500 mg/m^2 on Day 1 of Cycles 2-6. Chlorambucil: 10 milligrams per square meter per day (mg/m^2/day) oral administration (PO) on Days 1 to 7 of Cycles 1-6; 10 mg/m^2/day PO on Days 1 to 7 of Cycles 7-12, if applicable.
Period: Treatment Period
Arm/Group | Rituximab + Chlorambucil
Started | 100
Completed | 51
Not Completed | 49
Not completed — Adverse event/Serious adverse event | 25
Not completed — Physician Decision | 15
Not completed — Disease progression | 3
Not completed — Protocol Violation | 1
Not completed — Other | 5
Period: Follow-up Period
Arm/Group | Rituximab + Chlorambucil
Started | 98
Completed | 33
Not Completed | 65
Not completed — Adverse event/Serious adverse event | 1
Not completed — Disease progression | 57
Not completed — Lost to Follow-up | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised all participants recruited into the study and known to have received at least one dose of study treatment.
Groups:
- Rituximab + Chlorambucil: Participants received combination therapy of rituximab plus chlorambucil for first 6 cycles. Participants who did not achieve CR after Cycle 6 then received chlorambucil alone from Cycle 7 onwards until either they achieved a CR or for a maximum of 6 additional cycles. Rituximab: 375 mg/m^2 IV infusion on Day 1 of Cycle 1; 500 mg/m^2 on Day 1 of Cycles 2-6. Chlorambucil: 10 mg/m^2/day PO on Days 1 to 7 of Cycles 1-6; 10 mg/m^2/day PO on Days 1 to 7 of Cycles 7-12, if applicable.
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 56 days from the beginning of the last treatment cycle that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs as well as non-serious AEs.
Time Frame: First administration of study treatment up to 56 days after the beginning of the last treatment cycle (up to 365 days)
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 99

2. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of Clinical CR or Confirmed CR
Description: Clinical CR was achieved if all of the following criteria were met: a)Absence of lymphadenopathy (LD) by physical examination (PE) and Computed Tomography (CT) scan (all lymph nodes less than [<] 1.5 centimeters [cm] in diameter), b)No hepatomegaly (HM)/splenomegaly (SM) by PE/CT scan, c)Absence of B symptoms (unexplained fever greater than [>] 38 degrees [°] Centigrade [C], drenching night sweats/>10 percent [%] body weight loss in the last 6 months), d)Normal Complete Blood Count (CBC) (i. Leukocytes (Leuk) greater than or equal to [≥] 1.5×10^9 per liter (/L), ii. Platelets (Plat) >100×10^9/L, and iii. Haemoglobin (Hb) >11.0 grams per deciliter [g/dL]) and e)Once clinical, radiological and laboratory evaluations demonstrated CR, bone marrow (BM) biopsy and aspirate were performed 8 weeks later for confirmation; BM sample: normocellular for age, <30% of the cells being lymphocytes (Lym) and lymphoid nodules (LN) absent was considered as a confirmed CR.
Time Frame: Baseline until disease progression or death up to approximately 2.5 years (assessed at Baseline, Cycle 4 Day 1, Day 1 of Cycles 7-12, and thereafter every 3 months up to approximately 2.5 years; cycle length = 28 days)
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants
  Clinical CR | 37.0
  Confirmed CR | 10.0
  Clinical CR or Confirmed CR | 47.0

3. Secondary Outcome: Percentage of Participants With BOR of Partial Response (PR)
Description: PR was achieved if all of the following criteria were met: a)≥50% decrease in Lym count from the baseline value, b)≥50% reduction in LD by CT scan, c)≥50% reduction in size of liver/spleen by PE/CT scan and at least 1 of the following for a minimum of 8 weeks: i. Leuk ≥1.5×10^9/L or 50% improvement over baseline, ii. Plat >100×10^9/L or 50% improvement over baseline and iii. Hb >11.0 g/dL or 50% improvement over baseline without transfusion. Participants who fulfilled criteria for CR with persistent anemia/thrombocytopenia were considered in PRs. CR was achieved if all of the criteria were fulfilled for ≥8 weeks: a)Absence of LD by PE and CT scan, b)No HM/SM by PE/CT, c)Absence of B symptoms, d)Normal CBC, and e)BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent.
Time Frame: as for outcome 2
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 68.0

4. Secondary Outcome: Percentage of Participants With BOR of Nodular Partial Response (nPR)
Description: CR was achieved if all of the following criteria were met for ≥8 weeks: a)Absence of LD by PE and CT scan, b)No HM/SM by PE/CT scan, c)Absence of B symptoms, d)Normal CBC, and e)BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent. Participants with nPR were those who satisfied all of the CR criteria except for the BM, where LN could be identified histologically.
Time Frame: as for outcome 2
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 6.0

5. Secondary Outcome: Percentage of Participants With BOR of Progressive Disease (PD)
Description: PD is considered if 1 of the following criteria is met: a)≥50% increase in sum of the products of ≥2 lymph nodes compared to their smallest size (at least one ≥2 cm in diameter) or appearance of new lymph nodes/extranodal lesions, b)≥50% increase in the size of hepatosplenomegaly (HSM) as determined by PE/CT scan; appearance of palpable HM/SM that was not previously present, c)≥50% increase in the absolute number of circulating Lym to ≥5×10^9/L, d)Transformation to a more aggressive histology. Symptomatic deterioration (evident in clinical symptoms but not supported by tumor assessments), in such cases, the determination of clinical progression was based on symptomatic deterioration.
Time Frame: as for outcome 2
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 4.0

6. Secondary Outcome: Percentage of Participants With BOR of Stable Disease (SD)
Description: Participants without CR/PR or PD were considered having a tumor response of SD. CR: a) Absence of LD by PE and CT, b) No HM/SM by PE/CT, c) Absence of B symptoms, d) Normal CBC, and e) BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent. PR: a) ≥50% decrease in Lym count from baseline, b) ≥50% reduction in LD, c) ≥50% reduction in size of liver/spleen by PE/CT and ≥1 of the following for at least 8 weeks: i. Leuk ≥1.5×10^9/L or 50% improvement over baseline, ii. Plat >100×10^9/L or 50% improvement over baseline and iii. Hb >11.0 g/dL or 50% improvement over baseline without transfusion. PD: a) ≥50% increase in sum of the products of ≥2 lymph nodes compared to their smallest size or appearance of new lymph nodes/extranodal lesions, or b) ≥50% increase in the size of HSM; new appearance of palpable HM/SM, or c) ≥50% increase in the absolute number of circulating Lym to ≥5×10^9/L, or d) Transformation to a more aggressive histology.
Time Frame: as for outcome 2
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 11.0

7. Secondary Outcome: Percentage of Participants With Objective Response (CR or PR)
Description: Objective response was defined as a tumor response of CR or PR. CR was achieved if all of the criteria were met for ≥8 weeks: a)Absence of LD by PE and CT scan, b)No HM/SM by PE/CT scan, c)Absence of B symptoms, d)Normal CBC, and e)BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent. PR was achieved if all of the criteria were met: a)≥50% decrease in Lymp count from the baseline value, b)≥50% reduction in LD by CT scan, c)≥50% reduction in size of liver/spleen by PE/CT scan and at least 1 of the following for a minimum of 8 weeks: i. Leuk ≥1.5×10^9/L or 50% improvement over baseline, ii. Plat >100×10^9/L or 50% improvement over baseline and iii. Hb >11.0 g/dL or 50% improvement over baseline without transfusion. Participants who fulfilled criteria for CR with persistent anemia/thrombocytopenia were considered PRs.
Time Frame: as for outcome 2
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 84.0 [75.3 to 90.6]

8. Secondary Outcome: Percentage of Participant With Disease Progression or Death
Description: PD is considered if 1 of the following criteria is met: a)≥50% increase in sum of the products of ≥2 lymph nodes compared to their smallest size (at least one ≥2 cm in diameter) or appearance of new lymph nodes/extranodal lesions, b)≥50% increase in the size of HSM as determined by PE/CT scan; appearance of palpable HM/SM that was not previously present, c)≥50% increase in the absolute number of circulating Lym to ≥5×10^9/L, d)Transformation to a more aggressive histology. Symptomatic deterioration (evident in clinical symptoms but not supported by tumor assessments), in such cases, the determination of clinical progression was based on symptomatic deterioration.
Time Frame: as for outcome 2
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 68.0

9. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS was defined as the interval (in days) from trial treatment start date to earlier of the date of first tumor response assessment of PD or date of death by any cause. Participants who experienced none of these events or who were lost to follow-up at the time of analysis were censored on last date when they were assessed for tumor response. PD is considered if 1 of the following criteria is met: a)≥50% increase in sum of products of ≥2 lymph nodes compared to their smallest size (at least one ≥2 cm in diameter) or appearance of new lymph nodes/extranodal lesions, b)≥50% increase in the size of HSM as determined by PE/CT; appearance of palpable HM/SM that was not previously present, c)≥50% increase in the number of circulating Lym to ≥5×10^9/L, d)Transformation to a more aggressive histology. Symptomatic deterioration (evident in clinical symptoms but not supported by tumor assessments), in such cases, the determination of clinical progression was based on symptomatic deterioration.
Time Frame: as for outcome 2
Population: FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
days | 716.5 [500.0 to 784.0]

10. Secondary Outcome: Disease Free Survival (DFS) Time
Description: DFS time was defined as interval (in days) from first tumor response of CR to date of first tumor response of PD, or date of death by any cause. Participants who experienced none of these events or who were lost to follow-up at the time of analysis were censored on last date when they were assessed for tumor response. CR: a) Absence of LD by PE and CT, b) No HM/SM by PE/CT, c) Absence of B symptoms, d) Normal CBC, and e) BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent. PD: a) ≥50% increase in sum of the products of ≥2 lymph nodes compared to their smallest size or appearance of new lymph nodes/extranodal lesions, or b) ≥50% increase in the size of HSM; new appearance of palpable HM/SM, or c) ≥50% increase in the absolute number of circulating Lym to ≥5×10^9/L, or d) Transformation to a more aggressive histology.
Time Frame: as for outcome 2
Population: FAS population participants who achieved confirmed CR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 10
days | 855.0 [290.0 to 855.0]

11. Secondary Outcome: Duration of Response (DoR)
Description: DoR: defined as interval (in days) from first tumor response (of CR/PR/nPR) to earlier of date of PD/death. Participants without PD/death or who were lost to follow-up were censored. CR: a)Absence of LD by PE and CT, b)No HM/SM by PE/CT, c)Absence of B symptoms, d)Normal CBC, and e)BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent. PR: a)≥50% decrease in Lym count from baseline value, b)≥50% reduction in LD, c)≥50% reduction in size of liver/spleen by PE/CT scan and d)Leuk, Plat and Hb ≥1.5×10^9/L, >100×10^9/L and >11.0 g/dL, respectively or 50% improvement (of all the 3) over baseline value. nPR: participants who satisfied all of CR criteria except for BM, where LN could be identified. PD: a)≥50% increase in sum of the products of ≥2 lymph nodes or appearance of new lymph nodes/extranodal lesions, or b)≥50% increase in size of HSM; new appearance of palpable HM/SM, or c)≥50% increase in number of Lym, or d)Transformation to a more aggressive histology.
Time Frame: as for outcome 2
Population: FAS population participants who achieved confirmed CR, PR or nPR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 84
days | 645.0 [561.0 to 758.0]

12. Secondary Outcome: Percentage of Participants Who Died
Time Frame: as for outcome 2
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | 15.0

13. Secondary Outcome: Overall Survival (OS) Time
Description: This was defined as the interval (number of days) from the trial treatment start date to the date of death by any cause. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment.
Time Frame: as for outcome 2
Population: FAS.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 100
percentage of participants | NA [NA to NA] — Median and 95% confidence interval of OS time not available due to insufficient follow-up to allow estimation.

14. Secondary Outcome: Percentage of Participants Who Achieved Minimal Residual Disease (MRD) Negativity
Description: MRD negativity was defined by the absence of tumor cells in bone marrow, using 4-color flow cytometry. MRD was assessed in participants with a confirmed CR. CR was achieved if all of the following criteria were met for ≥8 weeks: a)Absence of LD by PE and CT scan, b)No HM/SM by PE/CT scan, c)Absence of B symptoms, d)Normal CBC, and e)BM biopsy: normocellular for age, <30% of the cells being Lym and LN absent.
Time Frame: as for outcome 2
Population: FAS population participants who achieved confirmed CR.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 10
percentage of participants | 0.0

15. Secondary Outcome: Mean Change From Baseline (CFB) in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Scores
Description: EORTC QLQ-C30: included global health status (GHS)/quality of life (QOL), functional scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Most questions used a 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used a 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores were averaged and transformed to 0-100 scale; a higher score for Global Qol/functional scales=better level of QoL/functioning, or a higher score for symptom scale=greater degree of symptoms.
Time Frame: Baseline, Day 1 of Cycles 5 and 11, end of follow-up (FU) (24 month [m] FU visit, up to approximately 3 years)
Population: FAS. Number of participants analyzed = number of participants evaluable for this outcome and n=number of participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Rituximab + Chlorambucil
Number analyzed (Participants) | 91
units on scale
  GHS/QoL score-baseline (n=91) | 65.7 (21.8)
  CFB in GHS/QoL Score-Cycle 5 (n=59) | 6.4 (21.7)
  CFB in GHS/QoL Score-Cycle 11 (n=40) | 6.2 (16.9)
  CFB in GHS/QoL Score-24m FU (n=17) | 2.0 (15.2)
  Physical functioning score-baseline (n=91) | 77.0 (22.3)
  CFB in physical functioning score-Cycle 5 (n=59) | 1.0 (15.3)
  CFB in physical functioning score-Cycle 11 (n=40) | 3.4 (22.0)
  CFB in physical functioning score-24m FU (n=17) | -2.0 (10.2)
  Role functioning score-baseline (n=91) | 73.4 (31.6)
  CFB in role functioning score-Cycle 5 (n=59) | 0.0 (28.9)
  CFB in role functioning score-Cycle 11 (n=40) | 3.8 (32.1)
  CFB in role functioning score-24m FU (n=17) | 3.9 (20.0)
  Emotional functioning score-baseline (n=91) | 82.5 (18.1)
  CFB in emotional functioning score-Cycle 5 (n=59) | 1.0 (16.5)
  CFB in emotional functioning score-Cycle 11 (n=40) | -0.1 (18.1)
  CFB in emotional functioning score-24m FU (n=17) | 0.5 (17.3)
  Cognitive functioning score-baseline (n=91) | 84.1 (19.1)
  CFB in cognitive functioning score-Cycle 5 (n=59) | -1.9 (15.4)
  CFB in cognitive functioning-Cycle 11 (n=40) | -0.4 (18.8)
  CFB in cognitive functioning-24m FU (n=17) | 5.2 (18.0)
  Social functioning score-baseline (n=91) | 82.2 (24.2)
  CFB in social functioning score-Cycle 5 (n=59) | 2.5 (22.5)
  CFB in social functioning score-Cycle 11 (n=40) | 0.0 (27.9)
  CFB in social functioning score-at 24m FU (n=17) | 5.2 (19.9)
  Fatigue score-baseline (n=91) | 33.4 (25.7)
  CFB in fatigue score-Cycle 5 (n=59) | -1.4 (24.9)
  CFB in fatigue score-Cycle 11 (n=40) | -6.1 (27.7)
  CFB in fatigue score-24m FU (n=17) | -5.6 (22.2)
  Nausea/vomiting score-baseline (n=91) | 6.2 (16.2)
  CFB in nausea/vomiting score-Cycle 5 (n=59) | 1.7 (20.9)
  CFB in nausea/vomiting score-Cycle 11 (n=40) | 0.4 (20.8)
  CFB in nausea/vomiting score-24m FU (n=17) | -2.9 (8.8)
  Pain score-baseline (n=91) | 17.8 (27.0)
  CFB in pain score-Cycle 5 (n=59) | -3.4 (28.8)
  CFB in pain score-Cycle 11 (n=40) | -1.3 (33.2)
  CFB in pain score-24m FU (n=17) | 0.0 (31.2)
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil; CFB in GHS/QoL statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.029, t-test, 2 sided
Statistical Analysis 2: Comparison: Rituximab + Chlorambucil; CFB in GHS/QoL statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.027, t-test, 2 sided
Statistical Analysis 3: Comparison: Rituximab + Chlorambucil; CFB in GHS/QoL statistical analysis at end of FU; Test type: Superiority or Other; p = 0.602, t-test, 2 sided
Statistical Analysis 4: Comparison: Rituximab + Chlorambucil; CFB in physical functioning statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.631, t-test, 2 sided
Statistical Analysis 5: Comparison: Rituximab + Chlorambucil; CFB in physical functioning statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.339, t-test, 2 sided
Statistical Analysis 6: Comparison: Rituximab + Chlorambucil; CFB in physical functioning statistical analysis at end of FU; Test type: Superiority or Other; p = 0.440, t-test, 2 sided
Statistical Analysis 7: Comparison: Rituximab + Chlorambucil; CFB in role functioning statistical analysis at Cycle 5; Test type: Superiority or Other; p = 1.000, t-test, 2 sided
Statistical Analysis 8: Comparison: Rituximab + Chlorambucil; CFB in role functioning statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.465, t-test, 2 sided
Statistical Analysis 9: Comparison: Rituximab + Chlorambucil; CFB in role functioning statistical analysis at end of FU; Test type: Superiority or Other; p = 0.431, t-test, 2 sided
Statistical Analysis 10: Comparison: Rituximab + Chlorambucil; CFB in emotional functioning statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.650, t-test, 2 sided
Statistical Analysis 11: Comparison: Rituximab + Chlorambucil; CFB in emotional functioning statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.980, t-test, 2 sided
Statistical Analysis 12: Comparison: Rituximab + Chlorambucil; CFB in emotional functioning statistical analysis at end of FU; Test type: Superiority or Other; p = 0.906, t-test, 2 sided
Statistical Analysis 13: Comparison: Rituximab + Chlorambucil; CFB in cognitive functioning statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.381, t-test, 2 sided
Statistical Analysis 14: Comparison: Rituximab + Chlorambucil; CFB in cognitive functioning statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.886, t-test, 2 sided
Statistical Analysis 15: Comparison: Rituximab + Chlorambucil; CFB in cognitive functioning statistical analysis at end of FU; Test type: Superiority or Other; p = 0.264, t-test, 2 sided
Statistical Analysis 16: Comparison: Rituximab + Chlorambucil; CFB in social functioning statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.424, t-test, 2 sided
Statistical Analysis 17: Comparison: Rituximab + Chlorambucil; CFB in social functioning statistical analysis at Cycle 11; Test type: Superiority or Other; p = 1.000, t-test, 2 sided
Statistical Analysis 18: Comparison: Rituximab + Chlorambucil; CFB in social functioning statistical analysis at end of FU; Test type: Superiority or Other; p = 0.312, t-test, 2 sided
Statistical Analysis 19: Comparison: Rituximab + Chlorambucil; CFB in fatigue statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.664, t-test, 2 sided
Statistical Analysis 20: Comparison: Rituximab + Chlorambucil; CFB in fatigue functioning statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.170, t-test, 2 sided
Statistical Analysis 21: Comparison: Rituximab + Chlorambucil; CFB in fatigue statistical analysis at end of FU; Test type: Superiority or Other; p = 0.318, t-test, 2 sided
Statistical Analysis 22: Comparison: Rituximab + Chlorambucil; CFB in Nausea/vomiting statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.536, t-test, 2 sided
Statistical Analysis 23: Comparison: Rituximab + Chlorambucil; CFB in nausea/vomiting statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.900, t-test, 2 sided
Statistical Analysis 24: Comparison: Rituximab + Chlorambucil; CFB in nausea/vomiting statistical analysis at end of FU; Test type: Superiority or Other; p = 0.188, t-test, 2 sided
Statistical Analysis 25: Comparison: Rituximab + Chlorambucil; CFB in pain statistical analysis at Cycle 5; Test type: Superiority or Other; p = 0.370, t-test, 2 sided
Statistical Analysis 26: Comparison: Rituximab + Chlorambucil; CFB in pain statistical analysis at Cycle 11; Test type: Superiority or Other; p = 0.813, t-test, 2 sided
Statistical Analysis 27: Comparison: Rituximab + Chlorambucil; CFB in pain statistical analysis at end of FU; Test type: Superiority or Other; p = 1.000, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: First administration of study treatment up to 56 days after the beginning of the last treatment cycle (up to 365 days)
Arm/Group | Rituximab + Chlorambucil
Serious Adverse Events (participants affected / at risk) | 39/100
Other Adverse Events (participants affected / at risk) | 97/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chlorambucil (N=100)
Neutropenic sepsis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Anal infection (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Encephalitis viral (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Infusion related reaction (General disorders) | 3
Pyrexia (General disorders) | 2
Oedema peripheral (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutropenic colitis (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Autonomic nervous system imbalance (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cytokine release syndrome (Immune system disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Staphylococcal indentification test positive (Investigations) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chlorambucil (N=100)
Anaemia (Blood and lymphatic system disorders) | 20
Leukopenia (Blood and lymphatic system disorders) | 23
Lymphopenia (Blood and lymphatic system disorders) | 41
Neutropenia (Blood and lymphatic system disorders) | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 19
Dyspepsia (Gastrointestinal disorders) | 8
Mouth ulceration (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 51
Vomiting (Gastrointestinal disorders) | 22
Chills (General disorders) | 17
Fatigue (General disorders) | 31
Infusion related reaction (General disorders) | 5
Mucosal inflammation (General disorders) | 6
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 27
Hypersensitivity (Immune system disorders) | 5
Cellulitis (Infections and infestations) | 5
Lower respiratory tract infection (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 5
Anorexia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 15
Headache (Nervous system disorders) | 15
Lethargy (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Drug eruption (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 13
Flushing (Vascular disorders) | 8
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.